CLINICAL TRIAL: NCT02315638
Title: Follow-up to Study Protocol B2801001, A Phase I/II, Open-Label Dose Escalation Study to Evaluate the Safety and Efficacy of Single Doses of TT-034 in Patients With Chronic Hepatitis C [CHC] Infection
Brief Title: Long-Term Follow-Up Safety Monitoring of Patients Dosed in the First-in-Man Phase I/II Study of TT-034.
Status: Terminated | Type: Observational
Why Stopped: Long term safety follow-up no longer required
Sponsor: Tacere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: B2801002
Record Dates: First submitted 2014-12-05; First posted 2014-12-12 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
Keywords: Adeno-associated viral vectors; Adeno-associated virus; AAV; AAV8; ddRNAi; shRNA; RNAi; Hepatitis; Chronic Hepatitis C; HCV; CHC; Genotype 1
MeSH Terms: conditions — Hepatitis C; Hepatitis; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected and archived for further testing, should future data suggest that it is clinically or scientifically indicated.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dosed subjects: There is no intervention. This is a observational study monitoring subjects that were dosed with TT-034 in the Tacere B2801001 study,

SUMMARY:
This is a long-term safety follow-up protocol for subjects who received TT-034 under the B2801001 protocol and consists of monitoring for at least 4.5 years.

DETAILED DESCRIPTION:
The main purpose of this follow-up study is to detect events suggestive of delayed adverse effects of the study drug by review of clinical histories and discussion with subjects to identify/elicit significant medical events, including but not limited to hematologic, malignant, autoimmune, neurologic, and hepatic events.

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment in Study B2801001 and dosing with TT-034
* An informed consent form for this study signed and dated by the subject or a legally acceptable representative

Exclusion Criteria:

* There are no specific exclusion criteria for this follow-up study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of subjects that were enrolled in Study B2801001 and who received a dose of TT-034.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-11; Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Long Term Safety as measured through an assessment of adverse events | 4.5 years
  The primary objective is to assess the long-term safety of TT-034 administered in subjects with CHC through an assessment of adverse events with a focus on hematologic, malignant, autoimmune, neurologic and hepatic events.

SECONDARY OUTCOMES:
Long Term Viral Load | 4.5 years
  The secondary objective is to monitor long-term HCV viral load, as available, of subjects who have received TT-034.

CONTACTS AND LOCATIONS:
Overall Officials: David Suhy, PhD, Study Director — Tacere Therapeutics, Inc.
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States